CLINICAL TRIAL: NCT01130298
Title: An Open-Label Study of Serum Testosterone Levels in Non-dosed Females After Secondary Exposure to Testosterone Gel 1.62% Applied to the Upper Arms and Shoulders and Use of a T-shirt Barrier
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S176.1.011
Record Dates: First submitted 2010-05-21; First posted 2010-05-26 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2011-06

CONDITIONS: Healthy
Keywords: testosterone,; Pharmacokinetics; replacement,; therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Testosterone Gel 1.62%

INTERVENTIONS:
Drug: Testosterone Gel 1.62% — 5 grams

SUMMARY:
Single-center, single dose, open-label study in healthy male and female volunteers to further characterize the transfer potential of Testosterone Gel 1.62% formulation.

DETAILED DESCRIPTION:
Single-center, single dose, open-label study in 12 healthy male and 12 healthy female volunteers to further characterize the transfer potential of Testosterone Gel 1.62% formulation.

ELIGIBILITY:
Inclusion Criteria

* BMI between 20-35 kg/m^2 inclusive.

Exclusion Criteria

* Males: history, current or suspected prostate or breast cancer.
* Females: pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration observed (Cmax) | Up to 5 days
  Maximum plasma concentration observed (Cmax) of total testosterone
Area Under the Plasma Concentration-time Curve (AUC) | Up to 5 days
  Area under the plasma concentration-time curve (AUC) of total testosterone
Average Plasma Concentration observed (Cav) | Up to 5 days
  Average Plasma Concentration observed (Cav) of total testosterone

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miller, PharmD, Study Director — Abbott

REFERENCES:
- [Result] Stahlman J, Britto M, Fitzpatrick S, McWhirter C, Testino SA, Brennan JJ, Zumbrunnen TL. Serum testosterone levels in non-dosed females after secondary exposure to 1.62% testosterone gel: effects of clothing barrier on testosterone absorption. Curr Med Res Opin. 2012 Feb;28(2):291-301. doi: 10.1185/03007995.2011.652732. Epub 2012 Jan 24. PMID 22188558